CLINICAL TRIAL: NCT01044771
Title: A Pilot Study to Evaluate the Effectiveness of a Tenofovir Raltegravir Switch in Resolving Tenofovir Induced Proteinuria in HIV Infected Individuals With Undetectable HIV Viral Loads
Brief Title: Pilot Study of Raltegravir Switch to Resolve Tenofovir Induced Proteinuria
Acronym: RALPIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metropolis Medical (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Fritz Bredeek, MD, PhD, President, Metropolis Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RALPIR
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections; Proteinuria
Keywords: HIV; Human immunodeficiency virus; tenofovir; viread; truvada; proteinuria
MeSH Terms: conditions — HIV Infections; Proteinuria; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- change from tenofovir to raltegravir (Other): Single arm study:
  Tenofovir containing nucleoside backbone changed over to raltegravir in all patients
  Interventions: Drug: change from tenofovir to raltegravir

INTERVENTIONS:
Drug: change from tenofovir to raltegravir — Change of the tenofovir based nucleoside part of the HIV regimen to raltegravir, 400mg BID
  Other Names: Isentress

SUMMARY:
The study is designed to evaluate the proportion of patients with tenofovir induced proteinuria that will resolve their proteinuria when the tenofovir containing nucleoside/nucleotide backbone is switched to a raltegravir backbone. Common HIV treatment regimens contain nucleoside/nucleotide combinations that may have long-term side effects including nephrotoxicity. Switching these backbones out for an integrase inhibitor based regimen has not been systematically evaluated.

Hypothesis: Proteinuria developing during treatment with tenofovir improves or resolves when tenofovir is switched out with raltegravir. Switching to a nuc- sparing regimen, containing raltegravir and a boosted protease inhibitor in patients without preexisting protease inhibitor mutations is safe and does not lead to virologic failure

DETAILED DESCRIPTION:
As described in the brief summary, this is a pilot study to evaluate for improvements in proteinuria when switched off from Tenofovir

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Ability to comply to protocol requirements
* On stable HAART for minimum of 12 weeks
* Evidence of TDF induced proteinuria
* No evidence of prior Protease inhibitor failure
* Treatment-naïve to integrase inhibitors
* VL<200 x 12 weeks (minimum of 2 viral load measurements)

Exclusion Criteria:

* Active Hepatitis B infection
* Proteinuria predating tenofovir use
* PRAMs on historic GT or PT
* Life expectancy less than 6 months
* Subjects with any ongoing AIDS defining illness
* Any condition which could compromise the safety of study subject
* Grade 3 or 4 lab abnormalities (excl. grade 3 bilirubin elevations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fritz Bredeek, MD, Principal Investigator — Metropolis Medical

RESULTS

PARTICIPANT FLOW:
Groups:
- Change From Tenofovir to Raltegravir: Single arm study:
  Tenofovir containing nucleoside backbone changed over to raltegravir in all patients Tenovovir 300mg was replaced with Raltegravir 400mg twice a day
Period: Overall Study
Arm/Group | Change From Tenofovir to Raltegravir
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HIV
Arm/Group | Change From Tenofovir to Raltegravir
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patients With Reduced or Resolved Proteinuria
Description: Measurement of Protein in Urine samples at end of study visit
Time Frame: 24 weeks
Measure: Number; unit: participants
Groups:
- Change From Tenofovir to Raltegravir: Single arm study:
  Tenofovir containing nucleoside backbone changed over to raltegravir in all patients
  change from tenofovir to raltegravir: Change of the tenofovir based nucleoside part of the HIV regimen to raltegravir, 400mg BID
Arm/Group | Change From Tenofovir to Raltegravir
Number analyzed (Participants) | 20
participants | 20

2. Secondary Outcome: Patients Without HIV Re-bound
Description: HIV Viral load blood test at week 24
Time Frame: 24 weeks
Population: Subjects entered with undetectable Viral Load and Proteinuria
Measure: Number; unit: participants
Groups:
- Viral Rebound: Every participant in the study switched to the investigational strategy
Arm/Group | Viral Rebound
Number analyzed (Participants) | 20
participants | 2

ADVERSE EVENTS:
Time Frame: during the study and 4 weeks after end of study
Arm/Group | Change From Tenofovir to Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No